CLINICAL TRIAL: NCT00941304
Title: A Double-Blind, Double-Dummy, Placebo- and Active Controlled Evaluation of the Efficacy, Safety and Tolerability of Buprenorphine HCl Buccal Film in the Treatment of Pain Associated With Third Molar Extraction
Brief Title: Study of Buprenorphine HCl Buccal Film in the Treatment of Dental Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUP-201
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Dental Pain
MeSH Terms: conditions — Toothache | interventions — Oxycodone; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Standard Opioid (Active Comparator): Oxycodone 5-mg oral capsule and 2 buccal placebo films
  Interventions: Drug: Oxycodone; Drug: Placebo Film
- High Dose buprenorphine HCl buccal film (Experimental): Buprenorphine HCl buccal film 0.5-mg modified formulation 1, buccal placebo film, and oral placebo capsule
  Interventions: Drug: Buprenorphine; Drug: Placebo Film; Drug: Placebo Capsule
- Mid Dose buprenorphine HCl buccal film (Experimental): Buprenorphine HCl buccal film 0.5-mg modified formulation 2, buccal placebo film, and oral placebo capsule
  Interventions: Drug: Buprenorphine; Drug: Placebo Film; Drug: Placebo Capsule
- Low Dose buprenorphine HCl buccal film (Experimental): Buprenorphine HCl buccal film 0.25-mg modified formulation 2, buccal placebo film, and oral placebo capsule
  Interventions: Drug: Buprenorphine; Drug: Placebo Film; Drug: Placebo Capsule
- Placebo (Placebo Comparator): Oral placebo capsule and 2 buccal placebo films
  Interventions: Drug: Placebo Film; Drug: Placebo Capsule

INTERVENTIONS:
Drug: Oxycodone — Single-dose of over-encapsulated oral 5-mg oxycodone capsule
  Other Names: Oxycodone capsule
  Arms: Standard Opioid
Drug: Buprenorphine — Single-dose of buprenorphine HCl buccal film
  Other Names: BEMA Buprenorphine; BELBUCA; Buprenorphine HCl buccal film; Buprenorphine HCl buccal soluble film
  Arms: High Dose buprenorphine HCl buccal film; Low Dose buprenorphine HCl buccal film; Mid Dose buprenorphine HCl buccal film
Drug: Placebo Film — Single-dose of placebo buccal film
  Other Names: Placebo; Placebo buccal film; BEMA placebo
Drug: Placebo Capsule — Single-dose of oral placebo capsule
  Other Names: Placebo; Oxycodone placebo
  Arms: High Dose buprenorphine HCl buccal film; Low Dose buprenorphine HCl buccal film; Mid Dose buprenorphine HCl buccal film; Placebo

SUMMARY:
The purpose of this study is to assess the activity of buprenorphine hydrochloride (HCl) buccal film in the treatment of dental pain.

ELIGIBILITY:
Inclusion Criteria:

* extraction of 2 or more third molars, at least 1 of which must be fully or partially impacted in mandibular bone
* males or non-pregnant females, aged 18 to 45 years
* good general health and capable of providing informed consent

Exclusion Criteria:

* history of substance abuse or dependence
* positive urine toxicology screen or alcohol breath test
* history of hypersensitivity to or allergy to any study drug
* donation of blood within prior 30 days
* use of analgesics, caffeine, sedatives, antidepressants, anticoagulant or antiplatelet agents within 24 hours

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Blum, MD, Study Director — BioDelivery Sciences International
Locations (3):
- United States (3):
  - Premier Research Group Limited, Austin, Texas
  - Donald P. Bandy, DDS, San Marcos, Texas
  - Premier Research Group Limited, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.25-mg Buprenorphine HCl Buccal Film, M2: Buprenorphine hydrochloride (HCl) buccal film 0.25-mg modified formulation 2, placebo buccal film, and placebo oral capsule
- 0.5-mg Buprenorphine HCl Buccal Film, M2: Buprenorphine HCl buccal film 0.5-mg modified formulation 2, placebo buccal film, and placebo oral capsule
- 0.5-mg Buprenorphine HCl Buccal Film, M1: Buprenorphine HCl buccal film 0.5-mg modified formulation 1, placebo buccal film, and placebo oral capsule
- Placebo: Placebo oral capsule and 2 placebo buccal films
- Oxycodone 5 mg: Oxycodone 5-mg oral capsule and 2 placebo buccal films
Period: Overall Study
Arm/Group | 0.25-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M1 | Placebo | Oxycodone 5 mg
Started | 31 | 30 | 31 | 30 | 31
Completed | 30 | 30 | 31 | 30 | 31
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis is based on Safety population; all subjects who received at least 1 dose of study drug.
Groups:
- 0.25-mg Buprenorphine HCl Buccal Film, M2: Buprenorphine HCl buccal film 0.25-mg modified formulation 2, placebo buccal film, and placebo oral capsule
- Total: Total of all reporting groups
Arm/Group | 0.25-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M1 | Placebo | Oxycodone 5 mg | Total
Number analyzed (Participants) | 31 | 30 | 31 | 30 | 31 | 153
Age, Continuous [Median (Full Range); unit: years] | 21.0 [18 to 30] | 21.0 [18 to 30] | 21.0 [18 to 27] | 22.0 [18 to 28] | 21.0 [18 to 29] | 21.0 [18 to 30]
Gender [Count of Participants; unit: Participants]
  Female | 22 | 20 | 20 | 18 | 16 | 96
  Male | 9 | 10 | 11 | 12 | 15 | 57

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference From Baseline to 8 Hours
Description: Time-weighted sum of pain intensity difference from baseline to 8 hours (SPID-8) where total score ranges from -80 (worst) to 80 (best) and a higher value indicates greater pain relief. Pain intensity was recorded using an 11-point numeric rating scale (NRS), where 0=none and 10=worst pain imaginable, in response to "What is your pain level at this time?"
Time Frame: Baseline, 8 hours
Population: Analysis based on intent-to-treat (ITT) population; all subjects who received study drug and provided at least 1 post-dose assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0.25-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M1 | Placebo | Oxycodone 5 mg
Number analyzed (Participants) | 31 | 30 | 31 | 30 | 31
units on a scale | 6.016 (19.9786) | 11.867 (20.7418) | 11.282 (22.9711) | 5.283 (17.6360) | 4.290 (14.8645)
Statistical Analysis 1: Comparison: 0.25-mg Buprenorphine HCl Buccal Film, M2 vs Placebo; Test type: Superiority or Other; p = .4739, ANCOVA; LS Mean Difference = 3.34, 95% CI 2-sided [-5.94 to 12.62]
Statistical Analysis 2: Comparison: 0.5-mg Buprenorphine HCl Buccal Film, M2 vs Placebo; Test type: Superiority or Other; p = .2183, ANCOVA; LS Mean Difference = 6.26, 95% CI 2-sided [-3.81 to 16.34]
Statistical Analysis 3: Comparison: 0.5-mg Buprenorphine HCl Buccal Film, M1 vs Placebo; Test type: Superiority or Other; p = .0809, ANCOVA; LS Mean Difference = 8.74, 95% CI 2-sided [-1.11 to 18.56]

2. Secondary Outcome: Total Pain Relief Over 8 Hours
Description: Time-weighted sum of total pain relief over 8 hours (TOPAR-8) where total score ranges from 0 (worst) to 32 (best) and higher values indicate greater pain relief. Pain relief (PAR) was recorded using a 5-point categorical rating scale, where 0=none, 1=a little, 2=some, 3=a lot, and 4=complete, in response to "How much relief have you had from your starting pain?"
Time Frame: 8 hours
Population: Analysis based on ITT population; all subjects who received study drug and provided at least 1 post-dose assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0.25-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M1 | Placebo | Oxycodone 5 mg
Number analyzed (Participants) | 31 | 30 | 31 | 30 | 31
units on a scale | 7.274 (8.7136) | 9.858 (9.3550) | 10.500 (9.9358) | 6.392 (8.6235) | 6.242 (6.6813)

3. Secondary Outcome: Sum of Pain Relief and Intensity Differences Over 8 Hours
Description: Time-weighted sum of PAR and pain intensity difference (PID) over 8 hours (SPRID-8) where total score ranges from -80 (worst) to 112 (best) and higher values indicate greater pain relief. PAR was recorded using a 5-point categorical rating scale, where 0=none, 1=a little, 2=some, 3=a lot, and 4=complete, in response to "How much relief have you had from your starting pain?" PID determined as the change from baseline pain intensity assessment. Pain intensity was recorded using an 11-point NRS, where 0=none and 10=worst pain imaginable, in response to "What is your pain level at this time?"
Time Frame: 8 hours
Population: Analysis based on ITT population; all subjects who received study drug and provided at least 1 post-dose assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0.25-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M1 | Placebo | Oxycodone 5 mg
Number analyzed (Participants) | 31 | 30 | 31 | 30 | 31
units on a scale | 13.290 (28.1677) | 21.725 (29.7031) | 21.782 (32.2047) | 11.675 (25.8038) | 10.532 (20.5848)

4. Secondary Outcome: Sum of Pain Relief and Intensity Differences Over 2 Hours
Description: Time-weighted sum of PAR and PID over 2 hours (SPRID-2) where total score ranges from 0 (worst) to 8 (best) and higher values indicate greater pain relief. PAR was recorded using a 5-point categorical rating scale, where 0=none, 1=a little, 2=some, 3=a lot, and 4=complete, in response to "How much relief have you had from your starting pain?" PID determined as the change from baseline pain intensity assessment. Pain intensity was recorded using an 11-point NRS, where 0=none and 10=worst pain imaginable, in response to "What is your pain level at this time?"
Time Frame: 2 hours
Population: Analysis based on ITT population; all subjects who received study drug and provided at least 1 post-dose assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0.25-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M1 | Placebo | Oxycodone 5 mg
Number analyzed (Participants) | 31 | 30 | 31 | 30 | 31
units on a scale | 0.339 (3.4896) | 1.533 (3.5718) | 1.056 (3.9769) | 0.850 (3.5505) | 1.484 (3.6009)

5. Secondary Outcome: Peak Pain Intensity Difference
Description: The maximum PID at any time following dosing determined from the change from baseline pain intensity assessment. Pain intensity was recorded using an 11-point NRS, where 0=none and 10=worst pain imaginable, in response to "What is your pain level at this time?"
Time Frame: 24 hours
Population: Analysis based on ITT population; all subjects who received study drug and provided at least 1 post-dose assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0.25-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M1 | Placebo | Oxycodone 5 mg
Number analyzed (Participants) | 31 | 30 | 31 | 30 | 31
units on a scale | 2.2 (3.50) | 2.9 (3.30) | 2.8 (3.35) | 1.5 (2.50) | 1.9 (2.61)

6. Secondary Outcome: Peak Pain Relief
Description: Maximum pain relief (PAR) at any time following dosing, recorded using a 5-point categorical rating scale, where 0=none, 1=a little, 2=some, 3=a lot, and 4=complete, in response to "How much relief have you had from your starting pain?"
Time Frame: 24 hours
Population: Analysis based on ITT population; all subjects who received study drug and provided at least 1 post-dose assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0.25-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M1 | Placebo | Oxycodone 5 mg
Number analyzed (Participants) | 31 | 30 | 31 | 30 | 31
units on a scale | 1.5 (1.59) | 1.8 (1.61) | 1.9 (1.51) | 1.1 (1.36) | 1.3 (1.33)

7. Secondary Outcome: Onset of Analgesia
Description: Time to onset of analgesia defined as median time to perceptible pain relief if confirmed by experiencing meaningful pain relief from time of study drug administration.
Time Frame: 8 hours
Population: Analysis based on ITT population; all subjects who received study drug and provided at least 1 post-dose assessment.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | 0.25-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M1 | Placebo | Oxycodone 5 mg
Number analyzed (Participants) | 31 | 30 | 31 | 30 | 31
hours | NA [3.083 to NA] — Median time to onset of analgesia and/or corresponding 95% confidence interval (CI) could not be determined as more than 50% of the subjects in treatment group failed to activate the stopwatch times within the protocol-specified 8-hour window. | 2.43 [0.617 to NA] — Median time to onset of analgesia and/or corresponding 95% confidence interval (CI) could not be determined as more than 50% of the subjects in treatment group failed to activate the stopwatch times within the protocol-specified 8-hour window. | NA [0.750 to NA] — Median time to onset of analgesia and/or corresponding 95% confidence interval (CI) could not be determined as more than 50% of the subjects in treatment group failed to activate the stopwatch times within the protocol-specified 8-hour window. | NA [NA to NA] — Median time to onset of analgesia and/or corresponding 95% confidence interval (CI) could not be determined as more than 50% of the subjects in treatment group failed to activate the stopwatch times within the protocol-specified 8-hour window. | NA [1.017 to NA] — Median time to onset of analgesia and/or corresponding 95% confidence interval (CI) could not be determined as more than 50% of the subjects in treatment group failed to activate the stopwatch times within the protocol-specified 8-hour window.

8. Secondary Outcome: Duration of Analgesia
Description: Duration of analgesia was the median time to use of rescue medication; earliest concomitant medication start time for medications identified as rescue medications from time of study drug administration.
Time Frame: 24 hours
Population: Analysis based on ITT population; all subjects who received study drug and provided at least 1 post-dose assessment.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | 0.25-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M1 | Placebo | Oxycodone 5 mg
Number analyzed (Participants) | 31 | 30 | 31 | 30 | 31
hours | 1.75 [1.667 to 5.083] | 2.62 [1.783 to 19.117] | 4.12 [2.067 to NA] — Corresponding 95% CI for duration of analgesia could not be determined as many subjects did not use rescue medication within 24 hours. | 1.69 [1.583 to 3.300] | 2.17 [1.683 to 2.750]

9. Secondary Outcome: Percentage of Participants Reporting a Global Rating of Study Drug as "Excellent"
Description: Subjects rated the global effectiveness of study drug as poor, fair, good, or excellent, in response to "Overall, how would you rate the study medication you received for pain?"
Time Frame: 8 hours and 24 hours
Population: Analysis based on ITT population; all subjects who received study drug and provided at least 1 post-dose assessment.
Measure: Number; unit: percentage of participants
Arm/Group | 0.25-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M1 | Placebo | Oxycodone 5 mg
Number analyzed (Participants) | 31 | 30 | 31 | 30 | 31
percentage of participants
  Excellent at 8 hours | 3.2 | 6.7 | 9.7 | 6.7 | 3.2
  Excellent at 24 hours | 9.7 | 13.3 | 12.9 | 3.3 | 0

10. Secondary Outcome: Percentage of Participants With "Excellent" Investigator Global Rating of Study Drug
Description: Investigators rated the global effectiveness of study drug as poor, fair, good, or excellent, in response to "Overall, how would you rate the study medication for this subject?"
Time Frame: 24 hours
Population: Analysis based on ITT population; all subjects who received study drug and provided at least 1 post-dose assessment.
Measure: Number; unit: percentage of participants
Arm/Group | 0.25-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M1 | Placebo | Oxycodone 5 mg
Number analyzed (Participants) | 31 | 30 | 31 | 30 | 31
percentage of participants | 6.5 | 13.3 | 12.9 | 3.3 | 0

11. Secondary Outcome: Change From Baseline in Cognitive Assessment Using CNS-VS
Description: Cognition assessed using computer-based CNS Vital Signs® neurocognitive function test (CNS-VS), including symbol digit coding, Stroop test, and shifting attention test to measure cognitive flexibility, executive functioning, processing speed, and reaction time(*). Scores are computed from raw score calculations using the data values of individual subtests. An asterisk denotes that "lower score is better", otherwise higher scores are better.
Time Frame: Baseline (screening), 2 hours 15 minutes postdose
Population: Analysis based on ITT population; all subjects who received study drug and provided at least 1 post-dose assessment.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | 0.25-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M1 | Placebo | Oxycodone 5 mg
Number analyzed (Participants) | 31 | 30 | 31 | 30 | 30
Score
  Cognitive flexibility | 5.9 (17.14) | 4.0 (18.93) | -3.2 (14.53) | 7.3 (10.81) | 2.1 (17.56)
  Executive functioning | 5.7 (17.35) | 4.1 (16.00) | -3.0 (13.49) | 7.2 (10.83) | 2.2 (17.19)
  Processing speed | -0.8 (7.64) | 0.8 (6.73) | -9.1 (14.48) | 2.8 (9.12) | 1.5 (9.63)
  Reaction time | 26.9 (79.82) | -19.5 (102.16) | 29.7 (157.55) | -3.5 (56.09) | -8.9 (61.13)

ADVERSE EVENTS:
Time Frame: From study drug administration (day 1) to follow-up visit (day 6 to 10)
Description: Analysis based on Safety population; all subjects who received any study drug
Arm/Group | 0.25-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M2 | 0.5-mg Buprenorphine HCl Buccal Film, M1 | Placebo | Oxycodone 5 mg
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/31 | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 9/31 | 18/30 | 25/31 | 3/30 | 6/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.25-mg Buprenorphine HCl Buccal Film, M2 (N=31) | 0.5-mg Buprenorphine HCl Buccal Film, M2 (N=30) | 0.5-mg Buprenorphine HCl Buccal Film, M1 (N=31) | Placebo (N=30) | Oxycodone 5 mg (N=31)
Nausea (Gastrointestinal disorders) | 6 (6) | 14 (14) | 20 (20) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 12 (12) | 16 (16) | 0 (0) | 0 (0)
Alveolar osteitis (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 5 (5) | 6 (7) | 13 (13) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other